CLINICAL TRIAL: NCT00123799
Title: A Phase II Study of Fluorodeoxyglucose (FluGlucoScan) in Patients With Breast Cancer: Correlation With Histologic Findings of Sentinel Node Biopsies and Axillary Dissection
Brief Title: Study of Fluorodeoxyglucose (FluGlucoScan) in Patients With Breast Cancer: Correlation With Histologic Findings of Sentinel Node Biopsies and Axillary Dissection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sufficient enrollment reached
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR-01-0057/DX-FDG-002/17097
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms
Keywords: positron emission tomography; fluorodeoxyglucose F18; sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Positron Emission Tomography Imaging

SUMMARY:
Breast cancer affects many women. One of the places to which it can spread is the lymph glands under the arm. The type of treatment offered to patients often will depend on whether those lymph glands have cancer in them or not. For this reason, a standard recommendation is that women with breast cancer have these lymph glands removed with surgery. This cancer causes side effects including numbness, pain, decreased ability to move the arm and arm swelling. A new type of surgery which looks only at the first gland that a cancer drains to (sentinel node biopsy) may help to avoid having to remove the glands under the arm. Also, a new way of imaging the glands under the arm called Positron Emission Tomography (PET) scanning may also give a better idea of the chance that these glands have cancer in them. This study is determining whether PET scans before surgery and sentinel node biopsy can decrease the need for a complete axillary dissection.

DETAILED DESCRIPTION:
1.0 Introduction

Breast cancer is the most common cancer in North American women. It is estimated that one in 8 American women will develop breast cancer during her lifetime. Surgical treatment has evolved from radical mastectomy to breast conservation, and systemic treatment has become increasingly important. The presence or absence of lymph node metastases is the most important prognostic factor used to determine type of systemic treatment necessary. Axillary dissection however, carries with it the risk of nerve injury, lymphedema, decreased arm motion and seroma formation. Clinical examination, ultrasound, CT scanning and MRI of the axilla are not sensitive or specific enough to eliminate the need for axillary dissection. Sentinel node biopsy (SNB) can predict the pathologic status of the axilla and theoretically could differentiate patients into those with positive node biopsies who require full dissection versus those who are negative and do not. Frozen section of the sentinel node is inaccurate and therefore SNB positive patients would require two surgical procedures. Positron Emission Tomography (PET) scanning of the axilla has been reported to have a high sensitivity and specificity and if used prior to surgery may guide the surgeon in determining the need for full axillary dissection versus SNB alone. PET scanning has also been reported to identify unsuspected distant metastases not found on standard staging examinations. This study will investigate the use of PET scanning in conjunction with SNB and results of both modalities will be correlated with histologic results of axillary dissection.

2.0 Objectives

There are no reports describing results of a similar study. By performing a properly constructed clinical trial in T1 - 3 N0 breast cancer patients, the question of whether PET scanning will make a difference to patient management can be answered. The hypothesis of this study is therefore, that a PET scan prior to surgery will facilitate staging both locally (axilla) and distant and will help the surgeon determine whether to do SNB or axillary dissection.

2.1 Primary Objective: To determine whether preoperative PET imaging combined with sentinel node biopsy can accurately identify nodal status. This would be most important in patients with a negative PET scan and negative sentinel nodes. If the combination of these tests was found to have a high negative predictive value for nodal metastases, full axillary dissection could be avoided.

2.2 Secondary Objectives:

* Assess pattern of lymph node drainage using lymphoscintigraphy.
* Assessment of size limitations of PET scanning in metastatic lymph nodes.
* Assessment of primary tumor size and evidence of multifocality as compared to preoperative imaging (mammography +/- ultrasound).
* The incidence of unsuspected distant metastases and frequency with which treatment was changed as a result of the PET scan would also be determined.

3.0 Materials and Methods

3.1 Patient Population: Pre and post menopausal women with clinical T1-3 N0 breast cancer are eligible. All will have biopsy proven breast carcinoma. Positive core or fine needle aspiration biopsies will be obtained in all patients. Core biopsies are preferred. Excisional biopsies are not allowed. Patients must not be pregnant or lactating and must not have had prior malignancy. Diabetic patients are ineligible. An informal survey of 8 patients from Calgary indicates that all 8 would be willing to travel to Edmonton for their PET scan. (Personal communication from Dr. Mews).

3.2 Preoperative Imaging: All patients will have preoperative mammography +/- ultrasound of the breast. Patients eligible for and consenting to the study will be referred to the Cross Cancer Institute by their surgeons and will have preoperative PET scanning. Imaging will be completed within seven days prior to surgery. Once a PET scanner becomes available in Calgary, the scans will be done there. Potential sites of distant metastases identified by PET scan will be imaged further and if necessary, possible biopsies will be obtained to confirm the diagnosis.

3.3 Surgery: Dr. Kelly Dabbs from Edmonton and Dr. Daphne Mew from Calgary will be the surgeons involved. They have proven experience in doing SNB's. At the time of surgery, sentinel node biopsy using both blue dye and colloid will be performed followed by level I/II axillary dissection. The patients may have either segmental resection or mastectomy.

3.4 Pathology: The sentinel node will be assessed by H&E as well as immunohistochemistry as per standard protocol. Measurements of primary tumor size, size of axillary metastases and size of in situ component will be documented. All pathology will be reported by Dr. J. Danyluk, Dr. R. Berendt and Dr. F. Alexander.

3.5 Outcome Analysis: Patients with positive axillary nodes on dissection and positive SNB and/or PET will be considered true positive (TP) for that modality. A negative axillary dissection and negative PET and/or SNB will identify the true negative (TN) group. A positive axillary dissection and negative PET and/or SNB will identify the false negative (FN) subgroup. A negative axillary dissection and positive PET and/or SNB will identify the false positive (FP) subgroup. Sensitivity (TP/TP + FN) and specificity (TN/TN + FP) will be determined. If patients do not have successful sentinel node surgery or PET scanning, they will be included in the analysis of the individual modality which was successful.

3.6 Statistics: In order to have an adequate number of node positive patients to test sensitivity an overall total of 240 patients is required. The proportion of patients who are node positive is estimated to be 0.35. A sample of 240 is expected to contain 84 node positive patients and the probability that at least 72 of the 240 patients are node positive is 0.95. The subsample of 72 node positive patients is sufficient to perform a one-sided test of equivalence for a target sensitivity of 0.80 and an allowable difference of 0.10 with significance level of 10% and power of 80%.The 168 node negative patients from the 240 total permit a one-sided test of equivalence for which the target specificity is 0.95 and the allowable difference is 0.05 with significance level of 5% and power of 90%.43

ELIGIBILITY:
Inclusion Criteria:

* Male or female. If female of child bearing potential and outside of the window of 10 days since the last menstrual period, a negative pregnancy test.
* Biopsy proven breast carcinoma (core biopsy or fine needle aspiration, although core biopsies are preferred.)
* Tumour size T1-3, N0 clinically
* All patients will have pre-operative mammography +/- ultrasound of the breast
* Age equal to or greater than 18 years
* Able and willing to follow instructions and comply with the protocol
* Provide written informed consent prior to participation in this study

Exclusion Criteria:

* Nursing or pregnant females
* Previous malignancy or diagnosis less than 10 (ten) years ago. Skin cancers (excluding malignant melanoma) and carcinoma in situ of the cervix are exceptions.
* Excisional biopsy of the tumour has been performed
* Age less than 18 years
* Patient has diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2004-06; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
to determine whether preoperative PET imaging combined with sentinel node biopsy can accurately identify axillary node status
to assess the size limitations of PET scanning in metastatic lymph nodes

SECONDARY OUTCOMES:
to determine the incidence of unsuspected distant metastases in patients with breast cancer
to determine the value of a delayed scan time of approximately three hours after the injection of 18F-FDG

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McEwan, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada